CLINICAL TRIAL: NCT03365193
Title: Retest prObability of Infectious ENDOCARDITIS for Appropriate Criteria Regarding Transesophageal ECHOcardiography in Tertiary Care Facilities
Brief Title: PRetest prObability of Infectious ENDOCARDITIS for Appropriate Criteria Regarding Transesophageal ECHOcardiography in Tertiary Care Facilities (PRO ENDOCARDITIS ECHO-Study)
Status: Completed | Type: Observational
Sponsor: University Hospital, Essen (Other)
Responsible Party: Principal Investigator, Amir Abbas Mahabadi, MD, coordinator cardiac trial unit, Principal Investigator, University Hospital, Essen
Other Study IDs: 17-7747-BO
Record Dates: First submitted 2017-12-01; First posted 2017-12-07 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2021-10

CONDITIONS: Infective Endocarditis
MeSH Terms: conditions — Endocarditis | interventions — Echocardiography, Transesophageal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Transesophageal Echocardiography — Standard transesophageal echocardiography will be performed as clinically indicated by treating physicians.

SUMMARY:
Infective endocarditis is a potentially lethal disease that has undergone major changes over the last decades. The Duke Criteria are recommended for evaluation of probability of presence of infective endocarditis by current ESC guidelines. However, since the introduction of Duke criteria in 1994, characteristics of patients presenting with potential infective endocarditis have substantially changed, especially in tertiary care facilities, towards a high proportion of patients with immune deficiency (caused by illness or medically induced), critically ill patients, patients with prosthetic valves and patients with long-lasting intensive care treatment. Likewise, with the increasing interventional therapy of structural heart disease and device implantation in older and multi-morbid patient cohorts, the frequency of endocarditis on prosthetic material and devices increased over the last decades. While Duke criteria overall misclassify a substantial proportion of patients with endocarditis, Duke criteria are difficult to apply in these patients because of lower sensitivity. Therefore, several modifications of the Duke criteria have been proposed. In addition, the uncertainty regarding potential infective endocarditis of treating physicians due to clinical characteristics of their patients leads to an increase in requests for transthoracic and transesophageal echocardiography, overcoming echocardiography laboratories. In the present study the investigators aim to identify (I) the precision of the Duke score in predicting presence of infective endocarditis in patients examined at the echocardiography laboratory of the West German Heart Center (II) determine characteristics, not including echocardiography that are associated with increased risk of infective endocarditis, justifying transesophageal echocardiography examination and (III) establish scoring algorithms to help treating physicians to assess the risk of endocarditis in severely diseased patient cohorts prior to echocardiography examinations and to avoid unnecessary echo exams.

ELIGIBILITY:
Inclusion Criteria:

* patients referred for echocardiographic assessment of suspected endocarditis

Exclusion Criteria:

* Unwillingness to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include patients with clinical indication for transesophageal echocardiography, as by decision of treating physicians.
Sampling Method: Probability Sample
Enrollment: 263 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2019-05-03 (Actual); Study Completion 2021-10-07 (Actual)

PRIMARY OUTCOMES:
Infective Endocarditis | From date of enrollment until hospital discharge, assessed up to 30 days
  Defined by an external clinical event committee

SECONDARY OUTCOMES:
Presence of signs of infective endocarditis on transesophageal echocardiography as defined by judgement of the examining physician. | At echocardiography examination.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Essen, Essen, North Rhine-Westphalia, Germany

REFERENCES:
- [Derived] Mahabadi AA, Mahmoud I, Dykun I, Totzeck M, Rath PM, Ruhparwar A, Buer J, Rassaf T. Diagnostic value of the modified Duke criteria in suspected infective endocarditis -The PRO-ENDOCARDITIS study. Int J Infect Dis. 2021 Mar;104:556-561. doi: 10.1016/j.ijid.2021.01.046. Epub 2021 Jan 27. PMID 33508475